CLINICAL TRIAL: NCT02199184
Title: Phase II Study of the Dose Adjusted EPOCH Regimen in Combination With Ofatumumab/Rituximab as Therapy for Patients With Newly Diagnosed or Relapsed/Refractory Burkitt Leukemia or Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Dose Adjusted EPOCH Regimen in Combination With Ofatumumab or Rituximab in Treating Patients With Newly Diagnosed or Relapsed or Refractory Burkitt Lymphoma or Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0123; NCI-2014-01707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0123 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: AIDS-Related Burkitt Lymphoma; Atypical Burkitt/Burkitt-Like Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent Acute Lymphoblastic Leukemia; Recurrent Burkitt Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Burkitt Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Etoposide; ofatumumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DA-EPOCH and ofatumumab or rituximab) (Experimental): Patients receive DA-EPOCH regimen comprising doxorubicin hydrochloride IV, vincristine sulfate IV, and etoposide IV continuously over 96 hours on days 1-4; cyclophosphamide IV over 1-2 hours on day 5; and prednisone PO BID on days 1-5. Patients also receive ofatumumab IV over 2 hours on days 1, 2, and 11 of cycle 1; on days 1 and 8 of cycles 2 and 4; and on days 1 and 11 of cycle 3 for a total of 9 injections. Patients may receive rituximab instead of ofatumumab if their insurance provider does not cover the cost of ofatumumab. Patients receive rituximab IV over 2 hours on days 1 and 11 of cycles 1 and 3 and on days 2 and 8 of cycles 2 and 4. Treatment repeats every 21-28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Ofatumumab; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2; Kesimpta
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well a dose adjusted regimen consisting of etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (EPOCH) works in combination with ofatumumab or rituximab in treating patients with Burkitt lymphoma that is newly diagnosed, or has returned after a period of improvement (relapsed), or has not responded to previous treatment (refractory) or relapsed or refractory acute lymphoblastic leukemia. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as ofatumumab and rituximab, may interfere with the ability of cancer cells to grow and spread. Giving more than one drug (combination chemotherapy) together with monoclonal antibody therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical efficacy of the combination of dose adjusted (DA)-EPOCH + ofatumumab in patients with newly diagnosed or relapsed/refractory Burkitt leukemia or relapsed/refractory acute lymphoblastic leukemia (ALL) defined by complete response rate.

SECONDARY OBJECTIVE:

I. To evaluate the safety of this combination, the overall survival and event-free survival rates.

OUTLINE:

Patients receive DA-EPOCH regimen comprising doxorubicin hydrochloride intravenously (IV), vincristine sulfate IV, and etoposide IV continuously over 96 hours on days 1-4; cyclophosphamide IV over 1-2 hours on day 5; and prednisone orally (PO) twice daily (BID) on days 1-5. Patients also receive ofatumumab IV over 2 hours on days 1, 2, and 11 of cycle 1; on days 1 and 8 of cycles 2 and 4; and on days 1 and 11 of cycle 3 for a total of 9 injections. Patients may receive rituximab instead of ofatumumab if their insurance provider does not cover the cost of ofatumumab. Patients receive rituximab IV over 2 hours on days 1 and 11 of cycles 1 and 3 and on days 2 and 8 of cycles 2 and 4. Treatment repeats every 21-28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-4 months for 1 year and then every 4-8 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Burkitt's or Burkitt-like leukemia/lymphoma, either previously untreated, or relapsed/refractory, or human immunodeficiency virus (HIV)-related; patients with double or triple hit high-grade leukemia/lymphoma are eligible also; patients HIV positive will be described and reported separately or relapsed/refractory acute lymphoblastic leukemia (ALL).
* Zubrod performance status =< 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Creatinine less than or equal to 2.0 mg/dL (unless considered tumor related)
* Bilirubin less than or equal to 2.0 mg/dL (unless considered tumor related)
* Adequate cardiac function defined as no history of clinically significant arrhythmia, or history of myocardial infarction (MI) within 3 months prior to study enrollment; cardiac function will be assessed by history and physical examination

Exclusion Criteria:

* Pregnant or nursing women
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 39 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Complete Remission: Normalization of the peripheral blood and bone marrow with 5% or less blasts in a normocellular or hypercellular marrow with a granulocyte count of 1 x 109/L or above and platelet count of 100 x 10^9/L or above. Complete resolution of all sites of extramedullary disease is required for CR.
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Number analyzed (Participants) | 14
Participants | 9

2. Secondary Outcome: Overall Survival Time
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 8 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Number analyzed (Participants) | 14
Months | 15.1 [1.8 to 95.3]

3. Secondary Outcome: Event-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 8 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Number analyzed (Participants) | 14
Months | 3.3 [0.6 to 67.0]

4. Secondary Outcome: Complete Response Duration
Description: Response date to loss of response or last follow up.
Time Frame: Up to 8 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
Number analyzed (Participants) | 14
Months | 10.0 [1.2 to 66.4]

ADVERSE EVENTS:
Time Frame: Up to 8 years.
Arm/Group | Treatment (DA-EPOCH and Ofatumumab or Rituximab)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (DA-EPOCH and Ofatumumab or Rituximab) (N=14)
Catheter Related Infection (Infections and infestations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (DA-EPOCH and Ofatumumab or Rituximab) (N=14)
mucositis (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
anemia (Blood and lymphatic system disorders) | 2 (2)
anorexia (Gastrointestinal disorders) | 2 (2)
Back pain (General disorders) | 1 (1)
Bilirubin increase (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Bone Pain) (Injury, poisoning and procedural complications) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increase (Investigations) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
dyspnea (Reproductive system and breast disorders) | 1 (1)
Edema (legs) (General disorders) | 1 (1)
Edema, limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Genital Edema (Reproductive system and breast disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
hemorrhoid (Gastrointestinal disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
neuropathy (Nervous system disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 2 (2)
Platelet count decrease (Investigations) | 4 (4)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell count decrease (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02199184/Prot_SAP_000.pdf